CLINICAL TRIAL: NCT04898907
Title: A Single Part, Four-Way Crossover, Randomized, Partially-Blinded Study to Evaluate the Effect of Intravenous ANG-3777 on Baseline-Adjusted QT/QTc Interval in the Fasted State in Healthy Male and Female Subjects
Brief Title: Study Developed to Evaluate the Effect of ANG-3777 on QT/QTc Interval
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Angion Biomedica Corp (Industry)
Collaborators: Quotient Sciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ANG3777-HV5-104
Record Dates: First submitted 2021-05-19; First posted 2021-05-24 (Actual); Last update posted 2021-06-01 (Actual); Status verified 2021-05

CONDITIONS: Healthy Volunteer
MeSH Terms: interventions — terevalefim; Saline Solution; Moxifloxacin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Partially blinded study. Patients are blinded as to treatment assignment. Care Provider, Investigator, and Outcomes Assessor will be blinded to ANG-3777 IV or saline IV, but Moxifloxacin Hydrochloride pill will be provided open label.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- ANG-3777 (Therapeutic Dose) (Experimental): Administered IV as a single dose on two occasions for 30 minutes on the morning of Day 1 of each treatment period (total of 4), following an 8 hour overnight fast. There will be a minimum washout of 3 days between each study drug administration.
  Interventions: Drug: ANG-3777 (Therapeutic Dose)
- Normal Saline (Placebo Comparator): The placebo will be administered as a single dose on separate occasions intravenously as 30-minute infusions on the morning of Day 1 of each treatment period (total of 4), following an 8 hour overnight fast. There will be a minimum washout of 3 days between each study drug administration.
  Interventions: Drug: Placebo
- Moxifloxacin Hydrochloride (Active Comparator): The comparator will be administered as a single dose oral Moxifloxacin Hydrochloride tablet (open-label), with a total of 240 mL of water. There will be a minimum washout of 3 days between each study drug administration.
  Interventions: Drug: Moxifloxacin Hydrochloride
- ANG-3777 (Supra-therapeutic Dose) (Experimental): Administered IV as a single dose on two occasions for 30 minutes on the morning of Day 1 of each treatment period (total of 4), following an 8 hour overnight fast. There will be a minimum washout of 3 days between each study drug administration.
  Interventions: Drug: ANG-3777 (Supra-therapeutic Dose)

INTERVENTIONS:
Drug: ANG-3777 (Therapeutic Dose) — Arms assigned to this intervention will receive 2 mg/kg, IV, Fasted
  Other Names: Hepatocyte growth factor mimetic
  Arms: ANG-3777 (Therapeutic Dose)
Drug: ANG-3777 (Supra-therapeutic Dose) — Arms assigned to this intervention will receive 6 mg/kg, IV, Fasted
  Other Names: Hepatocyte growth factor mimetic
  Arms: ANG-3777 (Supra-therapeutic Dose)
Drug: Placebo — Arms assigned to this intervention will receive normal saline, IV, Fasted
  Other Names: Normal Saline
  Arms: Normal Saline
Drug: Moxifloxacin Hydrochloride — Arms assigned to this intervention will receive 400 mg, Oral, Fasted
  Arms: Moxifloxacin Hydrochloride

SUMMARY:
The purpose of this study is to evaluate the effect of ANG-3777 on placebo-corrected change from baseline, QT/corrected QT (QTc) interval, following single intravenous (IV) doses in healthy volunteer adults.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy males or non-pregnant, non-lactating healthy females
2. Aged 18 to 55 years inclusive at the time of signing informed consent
3. Body mass index (BMI) of 18.0 to 32.0 kg/m2 as measured at screening
4. Weight ≥50 kg and ≤100 kg at screening and admission
5. Must be willing and able to comply with all study requirements
6. Must be able to understand a written informed consent, which must be obtained prior to initiation of study procedures
7. Must agree to use an adequate method of contraception

Exclusion Criteria:

1. Subjects who have received any IMP in a clinical research study within 5 half-lives or within 30 days prior to first dose. However, in no event, shall the time between last receipt of IMP and first dose be less than 30 days.
2. Subjects who are study site or sponsor employees, or are immediate family members of a study site or sponsor employee
3. Evidence of current SARS-CoV-2 infection
4. History of any drug or alcohol abuse in the past 2 years
5. Regular alcohol consumption in males >21 units per week and females >14 units per week (1 unit = 12 oz 1 bottle/can of beer, 1 oz 40% spirit, or 5 oz glass of wine)
6. A confirmed positive alcohol urine test at screening or admission
7. Current smokers and those who have smoked within the last 12 months or current users of e-cigarettes and nicotine replacement products and those who have used these products within the last 12 months
8. A confirmed positive urine cotinine test at screening or admission.
9. Positive drugs of abuse test result

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Estimated)
Dates: Start 2021-06 (Estimated); Primary Completion 2021-09 (Estimated); Study Completion 2021-09 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in corrected QT interval by Fridericia's formula for ANG-3777 at the therapeutic and supra-therapeutic dose levels compared to placebo | Day 1, Day 5, Day 9 and Day 13

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey Levy, MD, PhD, Principal Investigator — Quotient Sciences - Miami, Inc.
Locations (1):
- Quotient Sciences, Miami, Florida, United States